CLINICAL TRIAL: NCT00860067
Title: A Randomized, Double-Blind, Active Controlled Study to Evaluate the Immunogenicity of MEDI3250 in Adults 18 to 49 Years of Age
Brief Title: A Study to Evaluate the Immunogenicity of Quadrivalent LAIV in Adults 18 to 49 Years of Age
Acronym: MI-CP185
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Judith Falloon, M.D., MedImmune, LLC an affiliate of AstraZeneca AB
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-CP185
Record Dates: First submitted 2009-03-09; First posted 2009-03-11 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-11

CONDITIONS: Healthy or Stable Underlying Chronic Medical Condition
Keywords: influenza, FluMist, adults, vaccine
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Q/LAIV (MEDI3250) (Experimental): Q/LAIV (quadrivalent influenza vaccine) (MEDI3250) was supplied in the Becton Dickinson (BD) Accuspray device that delivers a 0.2 mL total volume intranasal dose divided into each nostril (ie, administered as 0.1 mL per nostril). Each 0.2 mL dose contained 10^7.0 ± 0.5 fluorescent focus units (FFU) of each of 4 temperature-sensitive, cold-adapted, attenuated, 6:2 reassortant influenza strains (A/H1N1 [A/South Dakota/6/2007], A/H3N2 [A/Uruguay/716/2007], B/Victoria [B/Malaysia/2506/2004], and B/Yamagata [B/Florida/4/2006]).
  Interventions: Biological: Q/LAIV (MEDI3250)
- FluMist/B/Yamagata (Active Comparator): FluMist/B/Yamagata (trivalent influenza vaccine) was supplied in the BD Accuspray device that delivers a 0.2 mL total volume intranasal dose divided into each nostril (ie, administered as 0.1 mL per nostril). Each 0.2 mL dose contained 10^7.0 ± 0.5 FFU of each of 3 temperature-sensitive, cold-adapted, attentuated, 6:2 reassortant influenza strains (A/H1N1 [A/South Dakota/6/2007], A/H3N2 [A/Uruguay/716/2007], and B/Yamagata [B/Florida/4/2006])a B strain of the Yamagata lineage.
  Interventions: Biological: FluMist/B/Yamagata
- FluMist/B/Victoria (Active Comparator): FluMist/B/Victoria(trivalent influenza vaccine) was supplied in the BD Accuspray device that delivers a 0.2 mL total volume intranasal dose divided into each nostril (ie, administered as 0.1 mL per nostril). Each 0.2 mL dose contained 10^7.0 ± 0.5 FFU of each of 3 temperature-sensitive, cold-adapted, attenuated, 6:2 reassortant influenza strains (A/H1N1 [A/South Dakota/6/2007], A/H3N2 [A/Uruguay/716/2007], and B/Victoria [B/Malaysia/2506/2004])a B strain of the Victoria lineage.
  Interventions: Biological: FluMist/B/Victoria

INTERVENTIONS:
Biological: Q/LAIV (MEDI3250) — 0.2 mL dose at Day 0
  Other Names: MEDI3250
  Arms: Q/LAIV (MEDI3250)
Biological: FluMist/B/Yamagata — 0.2 mL dose at Day 0
  Other Names: FluMist
  Arms: FluMist/B/Yamagata
Biological: FluMist/B/Victoria — 0.2 mL dose at Day 0
  Other Names: FluMist
  Arms: FluMist/B/Victoria

SUMMARY:
The objective of this study was to show that quadrivalent live attenuated influenza vaccine (Q/LAIV; MEDI3250) produced antibody levels similar to those produced by the commercial vaccine, FluMist.

DETAILED DESCRIPTION:
This randomized, double-blind, active controlled, multicenter study enrolled 1,800 subjects who were 18 to 49 years of age. Subjects were randomized by site in a 4:1:1 fashion to receive a single dose of Q/LAIV, trivalent FluMist containing an influenza B strain from the Yamagata lineage (FluMist/B/Yamagata), or trivalent FluMist containing an influenza B strain from the Victoria lineage (FluMist/B/Victoria). The study was conducted at multiple sites in the USA in the influenza off-season.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 to 49 years, inclusive, on the day of randomization (reached his or her eighteenth year birthday but not yet reached his or her 50th year birthday) at the time of the dose of blinded investigational product
* Written informed consent and any locally required authorization obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Females of child-bearing potential, (ie, unless surgically sterile [eg, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy], had a sterile male partner, was at least 1 year post-menopausal, or practiced abstinence) must have used an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, or use of a condom with spermicide by the sexual partner) for 30 days prior to the first dose of investigational product, and must have agreed to continue using such precautions for 60 days after the dose of investigational product. In addition, the subject must also have had a negative urine or blood pregnancy test at screening and, if screening and Day 0 did not occur on the same day, on the day of vaccination prior to randomization. Investigator judgment was required to assess a female subject's capability of pregnancy.
* Healthy by medical history and physical examination OR presence of stable underlying chronic medical condition for which hospitalization was not required in the previous year
* Able to complete follow-up period of 180 days post dose of vaccine as required by the protocol
* Subject available by telephone
* Able to understand and comply with the requirements of the protocol, as judged by the investigator

Exclusion Criteria:

* Acute illness or evidence of significant active infection at randomization
* Fever ≥ 100.4°F (38°C) at randomization
* History of asthma
* Any drug therapy from 15 days prior to randomization or expected drug therapy through 30 days post dose with the exception of contraceptives or chronic medications that were well tolerated and were not initiated and/or did not have a dosage change within 90 days of randomization.
* Previous medical history or evidence of an intercurrent illness that might have compromised the safety of the subject in the study
* Current or expected receipt of immunosuppressive medications (inhaled and topical corticosteroids were permitted) including corticosteroids (≥ 20 mg/day of prednisone equivalent given daily or on alternate days for ≥ 14 days) within a 30-day window around dose of investigational product Note: topical corticosteroids for uncomplicated dermatitis were permitted according to the judgment of the investigator; topical calcineurin inhibitors were permitted in accordance with their package insert at entry and during study participation.
* Receipt of immunoglobulin or blood products within 90 days before randomization into the study or expected receipt during study participation
* Receipt of any investigational drug therapy or standard vaccine within 30 days before the dose of investigational product in this study through 30 days after the dose of investigational product (use of licensed agents for indications not listed in the package insert was permitted)
* Any known immunosuppressive condition or immune deficiency disease including known or suspected infection with human immunodeficiency virus (HIV)
* History of allergic disease or reactions likely to be exacerbated by any component of the investigational product including allergy to eggs, egg proteins, gentamicin, or gelatin; or serious, life threatening, or severe reactions to previous influenza vaccinations
* History of Guillain-Barré syndrome
* Use of antiviral agents with activity against influenza virus (including amantadine, rimantadine, oseltamivir and zanamivir) within 30 days prior to dose of investigational product or anticipated use within 30 days after vaccination
* Known or suspected mitochondrial encephalomyopathy
* Lactating woman
* History of alcohol or drug abuse that, in the opinion of the investigator, would have affected the subject's safety or compliance with study
* Any condition that, in the opinion of the investigator, would have interfered with evaluation of the investigational product or interpretation of subject safety or study results
* Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1800 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Falloon, M.D., Study Director — MedImmune LLC
Locations (18):
- United States (18):
  - Benchmark Research, Sacramento, California
  - California Research Foundation, San Diego, California
  - Benchmark Research, San Francisco, California
  - University Clinical Research-Deland, LLC, DeLand, Florida
  - Pharmax Research Clinic, Inc, Miami, Florida
  - University Clinical Research, Inc, Pembroke Pines, Florida
  - Miami Research Associates, South Miami, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Kentucky Pediatric / Adult Research, Bardstown, Kentucky
  - The Center for Pharmaceutical Research, PC, Kansas City, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Rochester Clinical Research, Inc., Rochester, New York
  - Clinical Research Associates, Inc, Nashville, Tennessee
  - Benchmark Research, Austin, Texas
  - Benchmark Research, Fort Worth, Texas
  - Advanced Clinical Research, West Jordan, Utah

REFERENCES:
- [Background] Block SL, Yi T, Sheldon E, Dubovsky F, Falloon J. A randomized, double-blind noninferiority study of quadrivalent live attenuated influenza vaccine in adults. Vaccine. 2011 Nov 21;29(50):9391-7. doi: 10.1016/j.vaccine.2011.09.109. Epub 2011 Oct 6. PMID 21983154

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1,924 participants provided written informed consent and were screened for the study. Of these, 1,800 participants were randomized into the study at 18 sites in the USA from 23Mar2009 and 26Mar2009.
Pre-assignment Details: Participants who provided written informed consent and who met the eligibility criteria were randomized by site at a 4:1:1 ratio to receive Q/LAIV, FluMist/B/Yamagata, or FluMist/B/Victoria. The randomization incorporated a block design with a fixed block size of 6.
Groups:
- Q/LAIV (MEDI3250): Q/LAIV (quadrivalent influenza vaccine) (MEDI3250) was supplied in the Becton Dickinson (BD) Accuspray device that delivers a 0.2 mL total volume intranasal dose divided into each nostril (ie, administered as 0.1 mL per nostril). Each 0.2 mL dose contained 10^7.0 ± 0.5 fluorescent focus units (FFU) of each of 4 temperature sensitive, cold-adapted, attenuated, 6:2 reassortant influenza strains (A/H1N1 [A/South Dakota/6/2007], A/H3N2 [A/Uruguay/716/2007], B/Victoria [B/Malaysia/2506/2004], and B/Yamagata [B/Florida/4/2006]).
- FluMist/B/Yamagata: FluMist/B/Yamagata (trivalent influenza vaccine) was supplied in the BD Accuspray device that delivers a 0.2 mL total volume intranasal dose divided into each nostril (ie, administered as 0.1 mL per nostril). Each 0.2 mL dose contained 10^7.0 ± 0.5 FFU of each of 3 temperate sensitive, cold-adapted, attentuated, 6:2 reassortant influenza strains (A/H1N1 [A/South Dakota/6/2007], A/H3N2 [A/Uruguay/716/2007], and B/Yamagata [B/Florida/4/2006]).
- FluMist/B/Victoria: FluMist/B/Victoria(trivalent influenza vaccine) was supplied in the BD Accuspray device that delivers a 0.2 mL total volume intranasal dose divided into each nostril (ie, administered as 0.1 mL per nostril). Each 0.2 mL dose contained 10^7.0 ± 0.5 FFU of each of 3 temperature sensitive, cold-adapted, attenuated, 6:2 reassortant influenza strains (A/H1N1 [A/South Dakota/6/2007], A/H3N2 [A/Uruguay/716/2007], and B/Victoria [B/Malaysia/2506/2004]).
Period: Overall Study
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata | FluMist/B/Victoria
Started | 1200 | 299 | 301
Completed | 1149 | 290 | 292
Not Completed | 51 | 9 | 9
Not completed — Lost to Follow-up | 46 | 9 | 9
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata | FluMist/B/Victoria | Total
Number analyzed (Participants) | 1200 | 299 | 301 | 1800
Age Continuous [Mean (Standard Deviation); unit: years]
  Participants | 32.6 (9.2) | 32.8 (9.2) | 32.8 (9.2) | 32.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 658 | 165 | 171 | 994
  Male | 542 | 134 | 130 | 806
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 264 | 67 | 78 | 409
  Not Hispanic or Latino | 936 | 232 | 223 | 1391
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaskan Native | 5 | 1 | 4 | 10
  Asian | 11 | 2 | 2 | 15
  Black or African American | 249 | 66 | 61 | 376
  Native Hawaiian or Other Pacific Islander | 4 | 2 | 2 | 8
  White | 916 | 228 | 230 | 1374
  Other | 8 | 0 | 1 | 9
  Multiracial | 7 | 0 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 1200 | 299 | 301 | 1800

OUTCOME MEASURES:

1. Primary Outcome: The 4 Post-dose Strain-specific Serum Hemagglutination Inhibition (HAI) Antibody Geometric Mean Titers (GMT) in the Q/LAIV (MEDI3250) Arm Are Noninferior to Those in the Comparator FluMist Group.
Description: Noninferior immune response was defined as having the upper bound of the 2-sided 95% confidence intervals (CIs) for the HAI antibody GMT ratio (FluMist comparator divided by Q/LAIV) ≤ 1.5 for each of the 4 strains.
Time Frame: Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198; FY=299; FV=301;All FM=600), had post-dose HAI measurement (Q=1182; FY=292; FV=298; All FM=590), and had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1181; FY=292; FV=297; All FM=589).
Measure: Geometric Mean (Full Range); unit: geometric mean titer
Groups:
- All FluMist: All FluMist group for A/H1N1 and A/H3N2 strains, where data from both the FluMist/B/Yamagata arm and the FluMist/B/Victoria arm were combined.
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata | FluMist/B/Victoria | All FluMist
Number analyzed (Participants) | 1181 | 292 | 297 | 589
geometric mean titer
  A/H1N1 | 5.9 [2 to 1024] | NA [NA to NA] — The comparators for the GMT ratios for the primary endpoint were subjects in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains. | NA [NA to NA] — The comparators for the GMT ratios for the primary endpoint were subjects in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains. | 6.5 [2 to 512]
  A/H3N2 | 7.5 [2 to 2896] | NA [NA to NA] — The comparators for the GMT ratios for the primary endpoint were subjects in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains. | NA [NA to NA] — The comparators for the GMT ratios for the primary endpoint were subjects in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains. | 7.8 [2 to 2048]
  B/Yamagata | 51.2 [2 to 2048] | 56.4 [2 to 2048] | NA [NA to NA] — The comparators for the GMT ratios for the primary endpoint were subjects who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains. | NA [NA to NA] — The comparators for the GMT ratios for the primary endpoint were subjects who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains.
  B/Victoria | 36.5 [2 to 2896] | NA [NA to NA] — The comparators for the GMT ratios for the primary endpoint were subjects who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains. | 33.6 [2 to 1024] | NA [NA to NA] — The comparators for the GMT ratios for the primary endpoint were subjects who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains.
Statistical Analysis 1: Comparison: Q/LAIV (MEDI3250) vs All FluMist; A/H1N1: Noninferior immune response was assessed by evaluating the upper bound of the 2-sided 95% CI for the ratio of A/H1N1 GMTs for the specified comparison. Geometric mean titers for the A/H1N1 influenza antibody measurements were calculated as: GMT = antilog^e (mean [log^e x]) where x was the assay result and e was the natural logarithm; Test type: Non-Inferiority or Equivalence — The immune response of Q/LAIV was to be declared noninferior to that of trivalent FluMist if the upper bound of the 95% CI for post dose A/H1N1 GMT ratio was ≤ 1.5. This corresponded to the statistical hypothesis of: Ho: Rj > 1.5 for any j and Ha: Rj ≤ 1.5 for all j, where Rj was the A/H1N1 post-dose GMT ratio: (FluMist B/Yamagata A/H1N1 + FluMist B/Victoria A/H1N1) divided by Q/LAIV A/H1N1; Bootstrapping; Confidence intervals calculated based on bootstrapping method; Ratio of geometric mean = 1.09, 95% CI 2-sided [1.01 to 1.18]
Statistical Analysis 2: Comparison: Q/LAIV (MEDI3250) vs All FluMist; A/H3N2: Noninferior immune response was assessed by evaluating the upper bound of the 2-sided 95% CI for the ratio of A/H3N2 GMTs for the specified comparison. Geometric mean titers for the A/H3N2 influenza antibody measurements were calculated as: GMT = antilog^e (mean [log^e x]) where x was the assay result and e was the natural logarithm; Test type: Non-Inferiority or Equivalence — The immune response of Q/LAIV was to be declared noninferior to that of trivalent FluMist if the upper bound of the 95% CI for post dose A/H3N2 GMT ratio was ≤ 1.5. This corresponded to the statistical hypothesis of: Ho: Rj > 1.5 for any j and Ha: Rj ≤ 1.5 for all j, where Rj was the A/H3N2 post-dose GMT ratio: (FluMist B/Yamagata A/H3N2 + FluMist B/Victoria A/H3N2) divided by Q/LAIV A/H3N2; Bootstrapping; Confidence intervals calculated based on bootstrapping method; Ratio of geometric means = 1.05, 95% CI 2-sided [0.96 to 1.14]
Statistical Analysis 3: Comparison: Q/LAIV (MEDI3250) vs FluMist/B/Yamagata; Noninferior immune response was assessed by evaluating the upper bound of the 2-sided 95% CI for the ratio of B/Yamagata GMTs for the specified comparison. Geometric mean titers for the B/Yamagata influenza antibody measurements were calculated as: GMT = antilog^e (mean [log^e x]) where x was the assay result and e was the natural logarithm; Test type: Non-Inferiority or Equivalence — The immune response of Q/LAIV was to be declared noninferior to that of trivalent FluMist if the upper bound of the 95% CI for post dose B/Yamagata GMT ratio was ≤ 1.5. This corresponded to the statistical hypothesis of: Ho: Rj > 1.5 for any j and Ha: Rj ≤ 1.5 for all j, where Rj was the B/Yamagata post-dose GMT ratio: (FluMist B/Yamagata) divided by (Q/LAIV B/Yamagata); Bootstrapping; Confidence intervals calculated based on bootstrapping method; Ratio of geometric mean = 1.10, 95% CI 2-sided [0.97 to 1.25]
Statistical Analysis 4: Comparison: Q/LAIV (MEDI3250) vs FluMist/B/Victoria; Noninferior immune response was assessed by evaluating the upper bound of the 2-sided 95% CI for the ratio of B/Victoria GMTs for the specified comparison. Geometric mean titers for the B/Victoria influenza antibody measurements were calculated as: GMT = antilog^e (mean [log^e x]) where x was the assay result and e was the natural logarithm; Test type: Non-Inferiority or Equivalence — The immune response of Q/LAIV was to be declared noninferior to that of trivalent FluMist if the upper bound of the 95% CI for post dose B/Victoria GMT ratio was ≤ 1.5. This corresponded to the statistical hypothesis of: Ho: Rj > 1.5 for any j and Ha: Rj ≤ 1.5 for all j, where Rj was the B/Victoria post-dose GMT ratio: (FluMist B/Victoria) divided by (Q/LAIV B/Victoria); Bootstrapping; Confidence intervals were calculated based on bootstrapping method; Ratio of geometric means = 0.92, 95% CI 2-sided [0.82 to 1.03]

2. Secondary Outcome: The Number of Participants (Regardless of Serostatus) Within Each Treatment Arm Who Experience Strain-specific Seroresponse Post Dose.
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline.
Time Frame: Day 0 and Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198; FY=298; FV=300; All FM=598), had pre-dose and post-dose HAI measurement (Q=1181; FY=292; FV=298; All FM=599), and had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1180; FY=292; FV=297; All FM=589).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata | FluMist/B/Victoria | All FluMist
Number analyzed (Participants) | 1180 | 292 | 297 | 589
participants
  A/H1N1 | 61 | NA — The comparators for the seroresponse were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains. | NA — The comparators for the seroresponse were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains. | 31
  A/H3N2 | 59 | NA — The comparators for the seroresponse were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains. | NA — The comparators for the seroresponse were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains. | 25
  B/Yamagata | 118 | 30 | NA — The comparators for the seroresponse were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains. | NA — The comparators for the seroresponse were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains.
  B/Victoria | 145 | NA — The comparators for the seroresponse were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains. | 35 | NA — The comparators for the seroresponse were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains.

3. Secondary Outcome: The Number of Serosusceptible Participants Within Each Treatment Arm Who Experience A/H1N1 Strain-specific Seroresponse Post Dose.
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline. Participants with a baseline HAI titer <= 8 were considered to be serosusceptible for that strain.
Time Frame: Day 0 and Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198; All FM=600), had pre-dose and post-dose HAI measurement (Q=1181; All FM=590), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1180; All FM=589), and were serosusceptible to the strain (Q=889; All FM=429).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist
Number analyzed (Participants) | 889 | 429
participants | 59 | 30

4. Secondary Outcome: The Number of Serosusceptible Participants Within Each Treatment Arm Who Experience A/H3N2 Strain-specific Seroresponse Post Dose.
Description: as for outcome 3
Time Frame: Day 0 and Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198; All FM=600), had pre-dose and post-dose HAI measurement (Q=1181; All FM=590), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1180; All FM=589), and were serosusceptible to the strain (Q=807; All FM=393).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist
Number analyzed (Participants) | 807 | 393
participants | 53 | 25

5. Secondary Outcome: The Number of Serosusceptible Participants Within Each Treatment Arm Who Experience B/Yamagata Strain-specific Seroresponse Post Dose.
Description: as for outcome 3
Time Frame: Day 0 and Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198; FY=299), had pre-dose and post-dose HAI measurement (Q=1181; FY=292), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1180; FY=292), and were serosusceptible to the strain (Q=197; FY=43).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata
Number analyzed (Participants) | 197 | 43
participants | 66 | 17

6. Secondary Outcome: The Number of Serosusceptible Participants Within Each Treatment Arm Who Experience B/Victoria Strain-specific Seroresponse Post Dose.
Description: as for outcome 3
Time Frame: Day 0 and Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198; FV=301), had pre-dose and post-dose HAI measurement (Q=1181; FV=298), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1180; FV=297), and were serosusceptible to the strain (Q=250; FV=66).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Victoria
Number analyzed (Participants) | 250 | 66
participants | 92 | 28

7. Secondary Outcome: The Number of Seropositive Participants Within Each Treatment Arm Who Experience A/H1N1 Strain-specific Seroresponse Post Dose.
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline. Participants with a baseline HAI titer > 8 were considered to be seropositive for that strain.
Time Frame: Day 0 and Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198; All FM=600), had pre-dose and post-dose HAI measurement (Q=1181; All FM=590), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1180; All FM=589), and were seropositive to the strain (Q=291; All FM=160).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist
Number analyzed (Participants) | 291 | 160
participants | 2 | 1

8. Secondary Outcome: The Number of Seropositive Participants Within Each Treatment Arm Who Experience A/H3N2 Strain-specific Seroresponse Post Dose.
Description: as for outcome 7
Time Frame: Day 0 and Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198, AFM=600), had pre-dose and post-dose HAI measurement (Q=1181, AFM=590), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1180; All FM=589), and were seropositive to the strain (Q=373, All FM=196).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist
Number analyzed (Participants) | 373 | 196
participants | 6 | 0

9. Secondary Outcome: The Number of Seropositive Participants Within Each Treatment Arm Who Experience B/Yamagata Strain-specific Seroresponse Post Dose.
Description: as for outcome 7
Time Frame: Day 0 and Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198, FY=299), had pre-dose and post-dose HAI measurement (Q=1181, FY=292), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q1180; FY=292), and were seropositive to the strain (Q=983, FY=249).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata
Number analyzed (Participants) | 983 | 249
participants | 52 | 13

10. Secondary Outcome: The Number of Seropositive Participants Within Each Treatment Arm Who Experience B/Victoria Strain-specific Seroresponse Post Dose.
Description: as for outcome 7
Time Frame: Day 0 and Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198, FV=301), had pre-dose and post-dose HAI measurement (Q=1181, FV=298), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1180; FV=297), and were seropositive to the strain (Q=930, FV=231).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Victoria
Number analyzed (Participants) | 930 | 231
participants | 53 | 7

11. Secondary Outcome: The Number of Participants (Regardless of Serostatus) Within Each Treatment Arm Who Achieved a Strain-specific HAI Antibody Titer ≥ 32 Post Dose.
Time Frame: Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198; FY=299; FV=301; All FM=600,), had post-dose HAI measurement (Q=1182; FY=292; FV=298; All FM=290), and had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1181; FY=292; FV=298; All FM=590).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata | FluMist/B/Victoria | All FluMist
Number analyzed (Participants) | 1181 | 292 | 297 | 589
participants
  A/H1N1 | 189 | NA — The comparators were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains. | NA — The comparators were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains. | 100
  A/H3N2 | 250 | NA — The comparators were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains. | NA — The comparators were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains. | 133
  B/Yamagata | 881 | 226 | NA — The comparators were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains. | NA — The comparators were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains.
  B/Victoria | 771 | NA — The comparators were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains. | 191 | NA — The comparators were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains and participants who received FluMist with a matching B strain for B/Yamagata and B/Victoria strains.

12. Secondary Outcome: The Number of Serosusceptible Participants Within Each Treatment Arm Who Achieved a A/H1N1 Strain-specific HAI Antibody Titer ≥ 32 Post Dose.
Description: Participants with a strain-specific baseline HAI titer ≤ 8 were considered to be serosusceptible to that strain.
Time Frame: Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198, All FM=600), had post-dose HAI measurement (Q=1182; All FM=590), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1181, All FM=589), and were serosusceptible to the strain(Q=889, All FM=429).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist
Number analyzed (Participants) | 889 | 429
participants | 17 | 5

13. Secondary Outcome: The Number of Serosusceptible Participants Within Each Treatment Arm Who Achieved a A/H3N2 Strain-specific HAI Antibody Titer ≥ 32 Post Dose.
Description: Participants with a strain-specific baseline HAI titer ≤ 8 were considered to be serosusceptible to that strain.
Time Frame: Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198; All FM=600), had post-dose HAI measurement (Q=1181; All FM=590), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1181; All FM=589), and were serosusceptible to the strain (Q=807; All FM=393).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist
Number analyzed (Participants) | 807 | 393
participants | 18 | 11

14. Secondary Outcome: The Number of Serosusceptible Participants Within Each Treatment Arm Who Achieved a B/Yamagata Strain-specific HAI Antibody Titer ≥ 32 Post Dose.
Description: Participants with a strain-specific baseline HAI titer ≤ 8 were considered to be serosusceptible to that strain.
Time Frame: Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198, FY=299), had post-dose HAI measurement (Q=1181, FY=292), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1181; FY=292), and were serosusceptible to the strain (Q=197, FY=43).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata
Number analyzed (Participants) | 197 | 43
participants | 44 | 11

15. Secondary Outcome: The Number of Serosusceptible Participants Within Each Treatment Arm Who Achieved a B/Victoria Strain-specific HAI Antibody Titer ≥ 32 Post Dose.
Description: Participants with a strain-specific baseline HAI titer ≤ 8 were considered to be serosusceptible to that strain.
Time Frame: Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198; FV=301), had post-dose HAI measurement (Q=1181; FV=298), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1181; FV=297), and serosusceptible (Q=250; FV=66).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Victoria
Number analyzed (Participants) | 250 | 66
participants | 57 | 16

16. Secondary Outcome: The Number of Seropositive Participants Within Each Treatment Arm Who Achieved a A/H1N1 Strain-specific HAI Antibody Titer ≥ 32 Post Dose.
Description: Participants with a baseline HAI titer > 8 were considered to be seropositive for that strain.
Time Frame: Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198; All FM=600), had post-dose HAI measurement (Q=1181; All FM=590) and had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1181; All FM=589), and were seropositive to the strain (Q=291; All FM=160).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist
Number analyzed (Participants) | 291 | 160
participants | 172 | 95

17. Secondary Outcome: The Number of Seropositive Participants Within Each Treatment Arm Who Achieved a A/H3N2 Strain-specific HAI Antibody Titer ≥ 32 Post Dose.
Description: Participants with a baseline HAI titer > 8 were considered to be seropositive for that strain.
Time Frame: Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198; All FM=600), had post-dose HAI measurement (Q=1182; AFM=590), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1181; All FM=589), and were seropositive to the strain (Q=373; All FM=196).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist
Number analyzed (Participants) | 373 | 196
participants | 232 | 122

18. Secondary Outcome: The Number of Seropositive Participants Within Each Treatment Arm Who Achieved a B/Yamagata Strain-specific HAI Antibody Titer ≥ 32 Post Dose.
Description: Participants with a baseline HAI titer > 8 were considered to be seropositive for that strain.
Time Frame: Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198; FY=299), had post-dose HAI measurement (Q=1182; FY=292), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1181; FY=292), and were seropositive to the strain (Q=983; FY=249).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata
Number analyzed (Participants) | 983 | 249
participants | 837 | 215

19. Secondary Outcome: The Number of Seropositive Participants Within Each Treatment Arm Who Achieved a B/Victoria Strain-specific HAI Antibody Titer ≥ 32 Post Dose.
Description: Participants with a baseline HAI titer > 8 were considered to be seropositive for that strain.
Time Frame: Day 28-35
Population: Participants who received a full dose of investigational product (Q=1198; FV=301), had post-dose HAI measurement (Q=1182; FV=298), had no protocol deviation that could have interfered with the generation or interpretation of an immune response (Q=1181; FV=297), and were seropositive to the strain (Q=930; FV=231).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Victoria
Number analyzed (Participants) | 930 | 231
participants | 714 | 175

20. Secondary Outcome: The Number of Participants Experiencing Each Solicited Symptom From Administration of Investigational Product Through 14 Days Post Vaccination
Description: Solicited symptoms were fever ≥ 100.4°F (38.0°C), runny/stuffy nose, sore throat, cough, headache, generalized muscle aches, decreased activity level (lethargy) OR tiredness/weakness, decreased appetite. Collection of specific solicited symptoms (sore throat, headache, generalized muscle aches) was omitted when, according to the judgment of the investigator, the subject was too young to reliably report a particular symptom.
Time Frame: Days 0-14
Population: The Evaluable Safety Population for solicited symptoms included participants who received any investigational product (Q=1198; All FM=600) and for whom any follow-up solicited symptom safety data were recorded during the summarized period (Q=1197; All FM=597).
Measure: Number; unit: participants
Groups:
- All FluMist: Data from both the FluMist/B/Yamagata arm and the FluMist/B/Victoria arm were combined.
Arm/Group | Q/LAIV (MEDI3250) | All FluMist
Number analyzed (Participants) | 1197 | 597
participants
  Any solicited symptom | 713 | 358
  Fever ≥ 100.4°F | 16 | 9
  Fever ≥ 101.3°F | 9 | 2
  Fever ≥ 102.2°F | 4 | 1
  Fever ≥ 103.1°F | 1 | 1
  Fever ≥ 104.0°F | 0 | 0
  Fever ≥ 104.9°F | 0 | 0
  Runny/stuffy nose | 522 | 236
  Sore throat | 227 | 118
  Cough | 163 | 75
  Headache | 338 | 164
  Generalized muscle aches | 121 | 59
  Decreased activity level (lethargy) or tiredness | 211 | 106
  Decreased appetite | 77 | 32

21. Secondary Outcome: The Number of Participants Reporting Any Adverse Event From Administration of Investigational Product Through 28 Days Post Vaccination
Description: Any untoward medical occurrence in a patient or clinical investigation in a subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Time Frame: Days 0-28 post vaccination
Population: The Safety Population included participants who received any investigational product (Q=1198; All FM=600) and for whom any follow-up safety data were recorded (Q=1198; All FM=598).
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist
Number analyzed (Participants) | 1198 | 598
participants | 210 | 118

22. Secondary Outcome: Number of Participants Reporting Any Serious Adverse Event From Administration of Investigational Product Through 28 Days Post Vaccination
Description: Serious adverse events were those that resulted in death; were life-threatening; resulted in inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability or incapacity; were a birth defect in the offspring of a study participant; or were an important medical event that may not have resulted in death, threatened life, or required hospitalization but that, based on appropriate medical judgment, may have jeopardized the subject and may have required medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Days 0-28 post vaccination
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist
Number analyzed (Participants) | 1198 | 598
participants | 2 | 2

23. Secondary Outcome: Number of Participants Reporting Any Serious Adverse Event From Administration of Investigational Product Through 180 Days Post Vaccination
Description: as for outcome 22
Time Frame: Days 0-180 post vaccination
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist
Number analyzed (Participants) | 1198 | 598
participants | 12 | 6

24. Secondary Outcome: Number of Participants Reporting New Onset Chronic Diseases From Administration of Investigational Product Through 180 Days Post Vaccination
Description: An NOCD was a newly diagnosed medical condition that was of a chronic, ongoing nature and was assessed by the investigator as medically significant.
Time Frame: Days 0-180 post vaccination
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist
Number analyzed (Participants) | 1198 | 598
participants | 11 | 4

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from the time of investigational product administration (Day 0) through Day 28. Treatment emergent SAEs were collected from the time of investigational product administration (Day 0) through Day 180.
Arm/Group | Q/LAIV (MEDI3250) | All FluMist
Serious Adverse Events (participants affected / at risk) | 12/1198 | 6/598
Other Adverse Events (participants affected / at risk) | 102/1198 | 57/598
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q/LAIV (MEDI3250) (N=1198) | All FluMist (N=598)
ARTERIOSPASM CORONARY (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 2 (2) | 0 (0)
GAS GANGRENE (Infections and infestations) | 1 (1) | 0 (0)
LOBAR PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ILIUM FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TRAUMATIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q/LAIV (MEDI3250) (N=1198) | All FluMist (N=598)
DIARRHOEA (Gastrointestinal disorders) | 10 (10) | 6 (7)
NAUSEA (Gastrointestinal disorders) | 11 (11) | 6 (6)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 14 (14) | 8 (8)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
HEADACHE (Nervous system disorders) | 9 (9) | 7 (7)
COUGH (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 6 (6)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 4 (4)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 9 (9)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.